CLINICAL TRIAL: NCT01704391
Title: Haemodynamic Response to Aortic Surgery
Status: Completed | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Helene Korvenius Nedergaard, MD, Sygehus Lillebaelt
Other Study IDs: S-20110154
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Aortic Aneurysm, Abdominal; Aortic Diseases; Acute Kidney Injury
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Diseases; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples taken from urinary catheter. Centrifuged, supernatant frozen at -80 degrees C. Immunoassay analyzed at Roche modular P quantifying NGAL.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aortic aneurysm patients: 10 patients with a CT verified diagnosis of aortic aneurysm demanding open elective surgical correction with insertion of vascular prosthesis
- Aortic occlusive disease patients: 10 patients with CT verified aortic occlusive disease demanding open elective surgical correction with insertion of vascular prosthesis

SUMMARY:
Open elective abdominal aortic surgery is a high risk procedure involving clamping of the aorta. Indications include abdominal aortic aneurysm (AAA) or aortic occlusive disease (AOD) causing lower limb ischaemia.

These patients are often regarded as one entity in postoperative study settings. However, previous studies indicate that risk profiles, inflammatory activity, and haemodynamic capacity may differ between these groups. The first aim of this study was to evaluate postoperative ICU-requirements after open elective abdominal aortic surgery, hypothesising that AAA-patients had longer ICU-stays and needed more mechanical ventilation or acute dialysis than did patients with AOD.

The investigators see a relatively high incidence of postoperative acute kidney injury (AKI) following aortic surgery. Neutrophil Gelatinase Associated Lipocalcin (NGAL) may be useful in the early diagnosis of postopeative AKI. However, NGAL is also known as a marker of inflammatory activation. The ischaemia-reperfusion injury and subsequent inflammatory response to aortic cross clamping may per se induce a rise in NGAL despite intact renal function. Therefore NGAL may not be a reliable marker of AKI after AAS.

The second aim of this study is to describe the changes in NGAL after AAS in patients with and without postoperative dialysis-dependent AKI.

ELIGIBILITY:
Inclusion Criteria:

* CT verified aortic aneurysm or aortic occlusive disease

Exclusion Criteria:

* age<18 y
* contraindications to the use of oesophagus doppler monitor, eg mycosis, perforation, stenosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients sceduled for elective open operation for aortic aneurysm disease and 10 patients sceduled for elective open operation for aortic occlusive disease
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | 24 hours postoperatively
  Number of patients with an ICU LOS > 24 hours
Post-operative need for dialysis | 72 hours postoperatively
  Number of patients developing dialysis dependency during the first 72 hours postoperatively

SECONDARY OUTCOMES:
Hemodynamic peroperative changes in AAD vs AOD | After anaesthesia induction, 10 minutes after aortic cross-clamping, 10 minutes after reperfusion, end of surgery
  Stroke volume, cardiac index, systemic vasular resistance is recorded for AAD- and AOD patients at five time points during the operation using CardioQ, an oesophagus doppler monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Lillebaelt Hospital, Kolding Hospital, Kolding, Denmark